CLINICAL TRIAL: NCT00709007
Title: Evaluating the Role of Directly Administered Antiretroviral Therapy (DAART) in Conjunction With Opiate Substitution in Delivery of Highly Active Antiretroviral Therapy to HIV-1-infected Injecting Drug Users (IDUs) in Chennai, India
Brief Title: Directly Administered Antiretroviral Therapy (DAART) Among HIV-1infected Injecting Drug Users (IDUs) in Chennai, India
Acronym: DAART+
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No participants satisfied eligibility criteria and were enrolled into the study since July 2008.
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Gregory M Lucas, Johns Hopkins University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA018577-03S1 (NIH)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2009-03

CONDITIONS: HIV Infections; Heroin Dependence
MeSH Terms: conditions — HIV Infections; Heroin Dependence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAART (Experimental): Participants are observed taking HIV medications by study staff on days when they receive opioid agonist therapy (sub-lingual buprenorphine) at the clinic.
  Interventions: Behavioral: Directly Administered Antiretroviral Therapy (DAART)
- SAT (Active Comparator): Participants take their HIV medications on their own but visit the clinic for opioid agonist substitution therapy.
  Interventions: Behavioral: SAT

INTERVENTIONS:
Behavioral: Directly Administered Antiretroviral Therapy (DAART) — Participants are observed taking HIV medications by study staff on days when they receive opioid agonist therapy (sub-lingual buprenorphine) at the clinic.
  Arms: DAART
Behavioral: SAT — Participants take their HIV medications by themselves.
  Arms: SAT

SUMMARY:
Though the HIV epidemic in India is predominantly among heterosexual populations, it is estimated that there are approximately 1.1 million injection drug users (IDUs) in India with HIV prevalence as high as 64% among IDUs in certain cities. In April 2004, the government of India launched a free-antiretroviral therapy roll-out program aimed at initiating 100,000 persons on HAART. Similar guidelines are currently being followed for the delivery and choice of HAART for IDU and non-IDU populations. However, IDUs have certain issues that complicate the delivery of HAART that need to be addressed by delivery programs such as delayed access to care, poor perceived adherence, and more rapid disease progression. This proposal will assess the feasibility and effectiveness of directly administered antiretroviral therapy (DAART) in conjunction with opioid substitution as a mode of delivery of HAART to IDUs in Chennai, India. To evaluate this objective we will conduct a randomized controlled pilot study of DAART vs self-administered therapy (SAT) among 100 HIV-1 infected treatment naïve IDUs who are enrolled in an opioid substitution program in Chennai and compare the following outcomes between the two arms: Primary Endpoint: Proportion of participants with viral load (VL) <400 copies/ml at 24 and 48 weeks; Secondary Endpoints: (1) Incidence of mortality and AIDS-defining illnesses at 24 and 48 weeks, (2) Changes in absolute CD4+ count from baseline at 24 and 48 weeks, and (3) Incidence of antiretroviral drug resistance at 24 and 48 weeks. Intention-to-treat analyses will be used. The study objective is in line with the priority areas identified in the Indian National AIDS Control Program Phase III (NACP III) and the results of this study will help inform the government of India on appropriate modes of delivery of HAART to IDUs. This study will also be among the first studies to be conducted in India to evaluate two different modes of delivery of HAART to IDUs.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Provide written informed consent
3. Permanent residence should be less than or equal to 15 kms (9.5 miles) from the YRGCSAR clinic
4. Be an injection drug user (by self-report)
5. Satisfy criteria for opioid dependence as per the DSM-IV criteria (see Appendix)
6. Urine screening must test positive for presence of opioids
7. Documented evidence of HIV infection (double ELISA: Murex HIV-1.2.O, Abbott Murex, UK and Vironostika® HIV Uni-form II Ag/Ab, Biomérieux, The Netherlands)
8. Be ART naïve (by self-report)
9. If female of childbearing potential (all of the following)

   * Have a negative urine pregnancy test
   * Be willing to use barrier based or oral contraceptive for the duration of the study if sexually active.
10. Satisfy Indian National Guidelines for initiation of HAART (any of the following)

    * Absolute CD4+ count < 200 cells/ µl
    * AIDS-defining illness with any CD4+ count
    * Absolute CD4+ count between 200 - 350 cell/ µl with HIV-related symptoms

Exclusion Criteria:

1. Requires a liquid preparation of ART or ART needs to be dosed more than twice daily
2. Indicates an intention to migrate in the next 48 weeks
3. Clinical or radiological signs of active tuberculosis
4. Any medical or psychiatric condition that the study physician believes to be a contraindication to study participation.
5. Enrolled in another HIV treatment program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
HIV RNA < 400 copies/ml | 48 weeks

SECONDARY OUTCOMES:
Incidence of mortality and/or AIDS-defining illnesses | 48 weeks
Change in absolute CD4+ count from baseline | 48 weeks
Incidence of antiretroviral drug resistance | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Lucas, MD,PhD, Principal Investigator — Johns Hopkins University School of Medicine, USA
Locations (1):
- YR Gaitonde Centre for Substance Abuse-Related Research (YRGCSAR), Chennai, Tamil Nadu, India